CLINICAL TRIAL: NCT06137274
Title: Phase 2 Trial of Adaptive Radiotherapy Boost for Head and Neck Squamous Cell Carcinomas
Brief Title: Phase 2 Trial of Adaptive Radiotherapy Boost for HNSCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22313
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Carcinoma; Head and Neck Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Adaptive Radiotherapy treatment (Experimental): Patients will undergo adaptive radiotherapy boost for head/neck squamous cell carcinomas. A base conventional IMRT plan of 46-50Gy in 2 Gy to gross disease in the primary/nodes and 41.4-45 Gy in 1.8 Gy to the elective nodes per fraction will be utilized. The MR simulation will be utilized for boost treatment planning. Patients will receive their 6th fraction of the week on the adaptive platform treating the gross disease until completion of the base plan to 20 Gy in 2Gy daily fractions (10 fractions). Each ART treatment will be recontoured/replanned by the treating head/neck radiation oncologist as deemed clinically or dosimetrically necessary.
  Interventions: Radiation: Intensity-modulated radiotherapy; Other: Magnetic Resonance Guidance

INTERVENTIONS:
Radiation: Intensity-modulated radiotherapy — All patients will be treated with intensity-modulated radiotherapy (IMRT) plans.
  Other Names: IMRT
Other: Magnetic Resonance Guidance — All patients will undergo combined CT and/or MR simulation and will be treated with a sequential-boost technique.
  Other Names: View Ray

SUMMARY:
The purpose of the study is to determine if it is feasible to use magnetic resonance imaging (MRI) to adjust a portion of radiation therapy for patients with head and neck squamous cell carcinoma . The technique under study will be used to personalize the study treatment based on response, keeping all treatments within standard of care guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* ECOG performance status of 0, 1
* Patients with histologically or cytologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, nasopharynx, hypopharynx, larynx, or unknown primary in the neck.
* Patients with measurable disease, either at primary site or neck per RECIST 1.1.
* For patients planned to receive chemotherapy, adequate hematologic, hepatic and renal function as outlined in protocol.
* International normalized ratio of prothrombin time (INR) and prothrombin time (PT) within 28 days before randomization must be WNL for the lab. Patients who are therapeutically treated with an agent such as warfarin may participate if they are on a stable dose and no underlying abnormality in coagulation parameters exists per medical history.
* Negative serum pregnancy test within before starting study treatment in woman with childbearing potential.

Exclusion Criteria:

* Pregnancy or lactation
* Patients who have had prior radiotherapy to the head and neck or prior systemic therapy for the index cancer.
* Patients who had undergone definitive surgery for the index cancer.
* Patients with distant metastatic disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Improvement in Mean OAR Dose Reduction | Up to 15 months
  Feasibility of MR adaptive boost technique, as defined as achieving a reduction of mean OAR (parotids, submandibular glands, pharynx, oral cavity, tubarial glands, larynx, esophagus, and thyroid) doses greater than 7.5% compared to unadapted CT based plan. If 18 of 25 patients are meet the mean OAR criteria the approach will be considered feasible.

SECONDARY OUTCOMES:
Percentage of patients achieving a complete anatomic response | Up to 15 months
  Percentage of patients achieving a complete anatomic response by CT Neck and Chest and/or PET/CT will be tabulated. The 95% CI by the exact binomial distribution will be reported.
Percentage of patients achieving a complete metabolic response | Up to 15 months
  Percentage of patients achieving a complete metabolic response by CT Neck and Chest and/or PET/CT will be tabulated. The 95% CI by the exact binomial distribution will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: George Yang, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States